CLINICAL TRIAL: NCT04212169
Title: A Phase 2 Randomized, Double-blinded, Placebo-controlled Study to Evaluate the Efficacy and Safety of MEDI3506 in Adult Subjects With Moderate-to-severe Atopic Dermatitis
Brief Title: Efficacy and Safety of MEDI3506 in Adult Subjects With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9182C00001; 2019-003304-12 (EudraCT Number)
Record Dates: First submitted 2019-11-04; First posted 2019-12-26 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-08

CONDITIONS: Atopic Dermatitis
Keywords: MEDI3506; Safety; Efficacy; Atopic Dermatitis; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Intervention Model Description: Participants will be randomised to receive MEDI3506 dose 1, MEDI3506 Dose 2 or MEDI3506 dose 3 or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigation product only will be prepared and administered by unmasked personnel. All subjects will receive the same number of injections at each dose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- MEDI3506 at dose level 1 (Experimental): Participant will receive multiple doses of MEDI3506 at dose level 1.
  Interventions: Drug: MEDI3506
- MEDI3506 at dose level 2 (Experimental): Participant will receive multiple doses of MEDI3506 at dose level 2.
  Interventions: Drug: MEDI3506
- MEDI3506 at dose level 3 (Experimental): Participant will receive multiple doses of MEDI3506 at dose level 3.
  Interventions: Drug: MEDI3506
- Placebo (Placebo Comparator): Participant will receive multiple doses of Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MEDI3506 — multiple doses
  Arms: MEDI3506 at dose level 1; MEDI3506 at dose level 2; MEDI3506 at dose level 3
Drug: Placebo — multiple doses
  Arms: Placebo

SUMMARY:
This is a research study to determine the efficacy and safety of investigational drug MEDI3506 for the treatment of adult subjects with Atopic Dermatitis.

DETAILED DESCRIPTION:
This is a research study to determine the efficacy and safety of investigational drug MEDI3506 for the treatment of adult subjects with Atopic Dermatitis.

Each participant will be assigned randomly to a treatment arm, which could be different strengths of the active treatment or a placebo which does not contain active treatment. Both Participants and investigators will be masked to the treatment assignment.

Approximately 152 participants will take part in this study. There is a 4 weeks screening period to determine eligibility. After eligibility is confirmed, participants will receive investigational drug or placebo during the 16 weeks treatment period. This is then followed by an 8-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years inclusive at the time of consent.
* Body mass index between 19.0 and 40.0 kg/m2 inclusive.
* Documented history of chronic AD, for at least 1 year prior to screening Visit 1.
* Meets at minimum 1 of the criteria, as follows:

  * History of inadequate response to topical medications for AD
  * Subject intolerance to treatment with topical medications for AD, or
  * Topical medications are otherwise medically inadvisable
* AD that affects ≥ 10% of the body surface area (BSA).
* An EASI score of ≥ 12 at Visit 1 and ≥ 16 at Visit 3 (Day 1).
* An IGA score of ≥ 3.

Exclusion Criteria:

* Any active medical or psychiatric condition, or other reason, that would interfere with evaluation of the investigational product or interpretation of subject safety or study results.
* Any other clinically relevant abnormal findings from physical examination (including vital signs and electrocardiogram [ECG]) or from safety laboratory analysis.
* Active dermatologic conditions that might confound the diagnosis of AD or would interfere with the assessment of the skin.
* Known active allergic or irritant contact dermatitis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-09-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (37):
- United States (12):
  - Research Site, Birmingham, Alabama
  - Research Site, Santa Monica, California
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Charlotte, North Carolina
  - Research Site, Tulsa, Oklahoma
  - Research Site, Providence, Rhode Island
  - Research Site, Spartanburg, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, San Antonio, Texas
- Australia (4):
  - Research Site, Box Hill
  - Research Site, Carlton
  - Research Site, East Melbourne
  - Research Site, Fremantle
- Germany (4):
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Hamburg
  - Research Site, Mahlow
- Poland (6):
  - Research Site, Bialystok
  - Research Site, Kielce
  - Research Site, Lodz
  - Research Site, Poznan
  - Research Site, Skierniewice
  - Research Site, Wroclaw
- Spain (3):
  - Research Site, Alcobendas
  - Research Site, Leganés
  - Research Site, Seville
- United Kingdom (8):
  - Research Site, Corby
  - Research Site, High Wycombe
  - Research Site, Kenilworth
  - Research Site, Northwood
  - Research Site, Romford
  - Research Site, Shipley
  - Research Site, Sidcup
  - Research Site, Wokingham

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9182C00001&attachmentIdentifier=48b9bbe6-f0ed-437d-a775-dbb096d8d00a&fileName=d9182c00001-csp-amendment-9_Redacted_For_posting_Final.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9182C00001&attachmentIdentifier=8505791d-2be3-4bba-9073-9f92e0b31305&fileName=d9182c00001-sap-v3_Redacted_For_posting.pdf&versionIdentifier=
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9182C00001&attachmentIdentifier=d9a38987-1db3-4e15-a11c-7f4b627341b5&fileName=d9182c00001-study-synopsis_Redacted_For_posting.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Pooled Placebo
- MEDI3506 Dose 1: MEDI3506 Dose 1 was administered SC to participants once every 4 weeks for 16 weeks
- MEDI3506 Dose 2: MEDI3506 Dose 2 was administered SC to participants once every 4 weeks for 16 weeks
- MEDI3506 Dose 3: MEDI3506 Dose 3 was administered SC to participants once every 4 weeks for 16 weeks
Period: Overall Study
Arm/Group | Placebo | MEDI3506 Dose 1 | MEDI3506 Dose 2 | MEDI3506 Dose 3
Started | 56 | 19 | 18 | 55
Completed | 42 | 16 | 13 | 42
Not Completed | 14 | 3 | 5 | 13
Not completed — Adverse Event | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 10 | 2 | 5 | 7
Not completed — Other reason, unspecified | 3 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MEDI3506 Dose 1 | MEDI3506 Dose 2 | MEDI3506 Dose 3 | Total
Number analyzed (Participants) | 56 | 19 | 18 | 55 | 148
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.3 (11.4) | 28.7 (8.9) | 37.9 (14.3) | 34.6 (11.8) | 33.4 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 8 | 7 | 25 | 67
  Male | 29 | 11 | 11 | 30 | 81
Race/Ethnicity, Customized [Number; unit: Participants]
  AMERICAN INDIAN OR ALASKA NATIVE | 0 | 0 | 0 | 0 | 0
  ASIAN | 8 | 5 | 3 | 6 | 22
  BLACK OR AFRICAN AMERICAN | 1 | 1 | 2 | 2 | 6
  MULTIPLE CATEGORIES CHECKED | 1 | 0 | 1 | 0 | 2
  NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | 0 | 0 | 0 | 0 | 0
  OTHER | 0 | 0 | 1 | 2 | 3
  WHITE | 46 | 13 | 11 | 45 | 115
Region of Enrollment [Number; unit: Participants]
  USA | 6 | 0 | 3 | 7 | 16
  Australia | 0 | 0 | 1 | 1 | 2
  Germany | 5 | 1 | 3 | 2 | 11
  Spain | 7 | 0 | 0 | 5 | 12
  United Kingdom | 34 | 13 | 9 | 35 | 91
  Poland | 4 | 5 | 2 | 5 | 16
Eczema Area and Severity Index (EASI) score [Mean (Standard Deviation); unit: Scores on a scale] — Eczema Area and Severity Index (EASI) score is a composite score of area of involvement and severity score of 4 different body areas. The severity score is based on erythema, oedema/papulation, excoriation and lichenification of 4 body areas which are head, trunk, upper limbs and lower limbs. The score ranges between 0 to 72 points. Higher EASI score indicates more severe disease.
  Scores on a scale | 28.81 (8.90) | 28.94 (11.66) | 28.36 (11.87) | 32.30 (10.86) | 30.07 (10.43)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Week 16 in EASI Score
Description: The EASI evaluates 4 anatomic regions for severity and extent of key disease signs and focuses on the acute and chronic signs of inflammation (ie, erythema, edema, papulation, excoriation, and lichenification). The maximum score is 72, with higher values indicating more severe disease. Analysis was performed using mixed effect model for repeated measures and MCP-mod dose response model.
Time Frame: Week 16
Population: ITT population. Data after study withdrawal or use of rescue therapy was excluded.
Measure: Least Squares Mean (Standard Error); unit: Percentage of change from baseline
Arm/Group | Placebo | MEDI3506 Dose 1 | MEDI3506 Dose 2 | MEDI3506 Dose 3
Number analyzed (Participants) | 55 | 19 | 17 | 54
Percentage of change from baseline
  Percent change from baseline to Week 16 in EASI score analysed using MCP-mod dose response model | NA (NA) — No dose response model selected from the MCP-mod analysis because the dose response was absent | NA (NA) — No dose response model selected from the MCP-mod analysis because the dose response was absent | NA (NA) — No dose response model selected from the MCP-mod analysis because the dose response was absent | NA (NA) — No dose response model selected from the MCP-mod analysis because the dose response was absent
  Percent change from baseline to Week 16 in EASI score analysed using a repeated measures mixed model | -51.31 (5.214) | -50.03 (7.419) | -45.43 (8.402) | -53.02 (4.858)
Statistical Analysis 1: Comparison: MEDI3506 Dose 1; Test type: Superiority; p = 0.888, Mixed Models Analysis; Mean Difference (Final Values) = 1.27, 90% CI 2-sided [-13.67 to 16.22], Standard Error of Mean 8.981 — Differences less than 0 favours MEDI3506
Statistical Analysis 2: Comparison: MEDI3506 Dose 2; Test type: Superiority; p = 0.549, Mixed Models Analysis; Mean Difference (Final Values) = 5.87, 90% CI 2-sided [-10.36 to 22.10], Standard Error of Mean 9.756 — Differences less than 0 favours MEDI3506
Statistical Analysis 3: Comparison: MEDI3506 Dose 3; Test type: Superiority; p = 0.807, Mixed Models Analysis; Mean Difference (Final Values) = -1.72, 90% CI 2-sided [-13.38 to 9.95], Standard Error of Mean 7.014 — Differences less than 0 favours MEDI3506

2. Secondary Outcome: Percentage of Subjects Achieving a 90% Reduction From Baseline in EASI Score at Week 16
Description: To further assess the effects of MEDI3506 compared with placebo on AD disease severity, in adult subjects with moderate-to-severe AD. Responders are subjects who achieved at least 90% reduction from baseline in EASI score.
Time Frame: Week 16
Population: ITT population. Subjects who discontinued IP, withdrew from study or used rescue medication were considered as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI3506 Dose 1 | MEDI3506 Dose 2 | MEDI3506 Dose 3
Number analyzed (Participants) | 56 | 19 | 18 | 55
Participants | 0 | 0 | 1 | 3

3. Secondary Outcome: Percentage of Subjects Achieving a 75% Reduction From Baseline in EASI Score at Week 16
Description: To further assess the effects of MEDI3506 compared with placebo on AD disease severity, in adult subjects with moderate-to-severe AD. Responders are subjects who achieved at least 75% reduction from baseline in EASI score.
Time Frame: Week 16
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI3506 Dose 1 | MEDI3506 Dose 2 | MEDI3506 Dose 3
Number analyzed (Participants) | 56 | 19 | 18 | 55
Participants | 4 | 2 | 1 | 10
Statistical Analysis 1: Comparison: MEDI3506 Dose 1; Test type: Superiority; p = 0.6396, Fisher Exact; Odds Ratio (OR) = 1.53, 90% CI 2-sided [0.19 to 9.94] — Odds ratio greater than 1 favours MEDI3506
Statistical Analysis 2: Comparison: MEDI3506 Dose 2; Test type: Superiority; p = 0.9999, Fisher Exact; Odds Ratio (OR) = 0.76, 90% CI 2-sided [0.03 to 6.38] — Odds ratio greater than 1 favours MEDI3506
Statistical Analysis 3: Comparison: MEDI3506 Dose 3; Test type: Superiority; p = 0.0935, Regression, Logistic; Odds Ratio (OR) = 2.89, 90% CI 2-sided [0.91 to 10.49] — Odds ratio greater than 1 favours MEDI3506

4. Secondary Outcome: Percentage of Subjects Achieving a 50% Reduction From Baseline in EASI Score at Week 16
Description: To further assess the effects of MEDI3506 compared with placebo on AD disease severity, in adult subjects with moderate-to-severe AD. Responders are subjects who achieved at least 50% reduction from baseline in EASI score.
Time Frame: Week 16
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI3506 Dose 1 | MEDI3506 Dose 2 | MEDI3506 Dose 3
Number analyzed (Participants) | 56 | 19 | 18 | 55
Participants | 12 | 5 | 5 | 16

5. Secondary Outcome: Percentage of Subjects Achieving an IGA of 0 (Clear) or 1 (Almost Clear) With at Least a 2 Grade Reduction From Baseline Score at Week 16
Description: The IGA allows investigators to assess overall AD disease severity at 1 given time point and consists of a 5-point severity scale from clear to very severe disease (0 = clear, 1 = almost clear, 2 = mild disease, 3 = moderate disease, and 4 = severe disease).
Time Frame: Week 16
Population: ITT population. Subjects who discontinued IP, withdrew from the study, or required rescue therapy were considered as non responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI3506 Dose 1 | MEDI3506 Dose 2 | MEDI3506 Dose 3
Number analyzed (Participants) | 56 | 19 | 18 | 55
Participants
  IGA response rate at Week 16 | 1 | 1 | 0 | 5
  IGA response rate at Week 16 using MCP-Mod dose-response analysis | NA — No dose response model was selected from MCP-mod analysis due to logistic regression not converging | NA — No dose response model was selected from MCP-mod analysis due to logistic regression not converging | NA — No dose response model was selected from MCP-mod analysis due to logistic regression not converging | NA — No dose response model was selected from MCP-mod analysis due to logistic regression not converging
Statistical Analysis 1: Comparison: MEDI3506 Dose 1; Test type: Superiority; p = 0.4450, Fisher Exact; Odds Ratio (OR) = 3.06, 90% CI 2-sided [0.08 to 119.65] — Odds ratio greater than one favour MEDI3506
Statistical Analysis 2: Comparison: MEDI3506 Dose 2; Test type: Superiority; p = 0.9999, Fisher Exact; Odds Ratio (OR) = 0, 90% CI 2-sided [0.0 to 28.0] — Odds ratio greater than 1 favours MEDI3506
Statistical Analysis 3: Comparison: MEDI3506 Dose 3; Test type: Superiority; p = 0.1132, Fisher Exact; Odds Ratio (OR) = 5.50, 90% CI 2-sided [0.75 to 130.35] — Odds ratio greater than 1 favours MEDI3506

6. Secondary Outcome: Percentage of Subjects Achieving a Reduction of ≥ 3 From Baseline to Week 16 in Weekly Mean of Daily Peak Pruritus NRS
Description: Peak pruritus (ie, worst itch experienced in the previous 24 hours) assessed using an Numerical Rating Scale (NRS; 0 to 10) with 0 = no itch and 10 = worst imaginable itch. The daily assessments were summarised as a weekly mean.
Time Frame: Week 16
Population: ITT population. Subjects who withdrew from the study or required rescue therapy considered as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI3506 Dose 1 | MEDI3506 Dose 2 | MEDI3506 Dose 3
Number analyzed (Participants) | 56 | 19 | 18 | 55
Participants | 9 | 3 | 3 | 12

7. Secondary Outcome: Change From Baseline to Week 16 in Weekly Mean of Daily Peak Pruritus NRS
Description: as for outcome 6
Time Frame: Week 16
Population: ITT population, excluding missing data at baseline or week 16.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | MEDI3506 Dose 1 | MEDI3506 Dose 2 | MEDI3506 Dose 3
Number analyzed (Participants) | 55 | 19 | 18 | 55
Scores on a scale | -1.41 (0.356) | -1.06 (0.519) | -2.01 (0.595) | -2.24 (0.348)

8. Secondary Outcome: Change From Baseline to Week 16 in Weekly Mean of Daily Peak Skin Pain NRS
Description: Skin pain (ie, worst skin pain experienced in the previous 24 hours) assessed using an NRS (0 to 10) with 0 = no pain and 10 = worst imaginable pain. The daily assessments were summarised as a weekly mean.
Time Frame: Week 16
Population: ITT population, excluding missing data at baseline or week 16.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | MEDI3506 Dose 1 | MEDI3506 Dose 2 | MEDI3506 Dose 3
Number analyzed (Participants) | 41 | 16 | 12 | 40
Scores on a scale | -1.44 (2.39) | -1.66 (2.62) | -1.52 (1.61) | -1.63 (2.30)

9. Secondary Outcome: SCORAD: Percent Change From Baseline to Week 16
Description: SCORAD is a clinical tool for assessing the severity of AD that evaluates the extent and intensity of AD lesions, in addition to subjective symptoms. The maximum total score is 103, with higher values indicating more severe disease.
Time Frame: Week 16
Population: ITT population, excluding missing data at baseline or week 16.
Measure: Mean (Standard Deviation); unit: Percentage of change from baseline
Arm/Group | Placebo | MEDI3506 Dose 1 | MEDI3506 Dose 2 | MEDI3506 Dose 3
Number analyzed (Participants) | 35 | 15 | 12 | 40
Percentage of change from baseline | -31.79 (25.09) | -29.88 (23.14) | -36.22 (25.34) | -39.42 (25.44)

10. Secondary Outcome: Change From Baseline to Week 16 in Percentage Body Surface Area (BSA) Affected by AD
Description: Change in percentage of body surface area (BSA) affected by AD from baseline at week 16.
Time Frame: Week 16
Population: ITT population, excluding missing data at baseline or week 16.
Measure: Mean (Standard Deviation); unit: Percentage of body surface area
Arm/Group | Placebo | MEDI3506 Dose 1 | MEDI3506 Dose 2 | MEDI3506 Dose 3
Number analyzed (Participants) | 37 | 15 | 13 | 40
Percentage of body surface area | -17.81 (17.09) | -11.07 (10.92) | -9.46 (13.23) | -23.13 (19.35)

11. Secondary Outcome: Change From Baseline to Week 16 in DLQI
Description: The Dermatology Life Quality Index (DLQI) is a 10-item, patient- completed, health-related quality of life assessment of dermatology conditions with a recall period of 1 week. Each item is scored on a 4-point Likert scale with 0 = not at all ⁄not relevant, 1 = a little, 2 = a lot, and 3 = very much. The score from each item is summed, and the maximum total score is 30 while the minimum score is 0. Higher score means highest (adverse) effect on participant's life.
Time Frame: Week 16
Population: ITT population, excluding missing data at baseline or week 16.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Placebo | MEDI3506 Dose 1 | MEDI3506 Dose 2 | MEDI3506 Dose 3
Number analyzed (Participants) | 38 | 15 | 12 | 40
Scores on scale | -2.9 (5.3) | -2.1 (6.5) | -2.4 (4.9) | -2.7 (4.9)

12. Secondary Outcome: Patient Description of Atopic Dermatitis or Eczema From Patient Global Impression of Severity at Week 16
Description: The Patient Global Impression of Severity (PGI-S) is a tool that allows patients to rate the severity of a condition over the past 7 days with response options of "No symptoms", "Very mild", "Mild", "Moderate", "Severe" and "Very severe".
Time Frame: Week 16
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI3506 Dose 1 | MEDI3506 Dose 2 | MEDI3506 Dose 3
Number analyzed (Participants) | 56 | 19 | 18 | 55
Participants
  No symptoms | 1 | 0 | 1 | 1
  Very mild | 5 | 0 | 5 | 10
  Mild | 9 | 4 | 2 | 8
  Moderate | 11 | 5 | 1 | 14
  Severe | 11 | 4 | 2 | 6
  Very severe | 1 | 2 | 1 | 1
  Missing data | 18 | 4 | 6 | 15

13. Secondary Outcome: Change From Baseline to Week 16 in POEM
Description: The Patient-Oriented Eczema Measure (POEM) is a 7-item questionnaire for assessing disease symptoms including dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping occurring in the past week. Each item is scored on a 5-point scale with 0 = no days, 1 = 1 to 2 days, 2 = 3 to 4 days, 3 = 5 to 6 days, and 4 = every day. The total POEM score is calculated by summing the score of each item resulting in a maximum of 28 and a minimum of 0, with higher values indicating severe disease
Time Frame: Week 16
Population: ITT population, excluding missing data at baseline or week 16.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Placebo | MEDI3506 Dose 1 | MEDI3506 Dose 2 | MEDI3506 Dose 3
Number analyzed (Participants) | 38 | 15 | 12 | 40
Scores on scale | -5.4 (7.9) | -2.5 (4.8) | -3.7 (8.7) | -6.3 (6.9)

14. Secondary Outcome: Change From Baseline to Week 16 in 5-D Itch
Description: The 5-D Itch Scale is a questionnaire consisting of 5 items used specifically to measure the course of itch by asking for the degree, duration, disability and distribution of the pruritus within the last 2 weeks. The scores from each item are summed, with maximum score of 25 and minimum score of 5. Higher score represent worse outcome
Time Frame: Week 16
Population: ITT population, excluding missing data at baseline or week 16.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Placebo | MEDI3506 Dose 1 | MEDI3506 Dose 2 | MEDI3506 Dose 3
Number analyzed (Participants) | 38 | 15 | 12 | 40
Scores on scale | -3.0 (4.9) | -3.0 (2.6) | -3.8 (3.4) | -4.0 (5.1)

15. Secondary Outcome: Occurrence of Adverse Events
Description: To assess the safety and tolerability of MEDI3506 compared with placebo, in adult subjects with moderate-to-severe AD.
Time Frame: up to 24 weeks
Population: As-treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI3506 Dose 1 | MEDI3506 Dose 2 | MEDI3506 Dose 3
Number analyzed (Participants) | 56 | 19 | 18 | 55
Participants
  At least one adverse event | 37 | 9 | 14 | 32
  At least one investigational product related event | 7 | 3 | 7 | 8
  At least one event of ≥ grade 3 severity | 7 | 2 | 2 | 5
  At least one serious event | 2 | 0 | 2 | 1
  At least one investigational product related serious event | 0 | 0 | 1 | 0

16. Secondary Outcome: Oral or Tympanic Temperature Taken During Vital Signs Assessment
Description: Collectively with other vital signs assessment are used to assess the safety and tolerability of MEDI3506 compared with placebo, in adult subjects with moderate-to-severe AD.
Time Frame: Baseline, week 16 and week 24
Population: As-treated population
Measure: Mean (Standard Deviation); unit: degrees C
Arm/Group | Placebo | MEDI3506 Dose 1 | MEDI3506 Dose 2 | MEDI3506 Dose 3
Number analyzed (Participants) | 56 | 19 | 18 | 55
degrees C
  Baseline | 36.46 (0.35) | 36.43 (0.52) | 36.41 (0.43) | 36.52 (0.39)
  Week 16: number analyzed (Participants) | 56 | 15 | 13 | 42
  Week 16 | 36.49 (0.36) | 36.71 (0.41) | 36.50 (0.32) | 36.47 (0.39)
  Week 24: number analyzed (Participants) | 56 | 15 | 13 | 40
  Week 24 | 36.44 (0.43) | 36.63 (0.50) | 36.55 (0.42) | 36.51 (0.37)

17. Secondary Outcome: Systolic Blood Pressure Taken During Vital Signs Assessment
Description: as for outcome 16
Time Frame: Baseline, week 16 and week 24
Population: As-treated population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | MEDI3506 Dose 1 | MEDI3506 Dose 2 | MEDI3506 Dose 3
Number analyzed (Participants) | 56 | 19 | 18 | 55
mmHg
  Baseline | 117.7 (12.9) | 119.3 (9.2) | 123.8 (9.9) | 121.5 (12.5)
  Week 16: number analyzed (Participants) | 56 | 15 | 13 | 42
  Week 16 | 117.8 (9.6) | 117.3 (7.2) | 120.7 (13.6) | 119.8 (10.6)
  Week 24: number analyzed (Participants) | 56 | 16 | 13 | 40
  Week 24 | 118.9 (11.1) | 117.6 (11.4) | 120.1 (15.1) | 120.6 (12.1)

18. Secondary Outcome: Heart Rate Taken During Vital Signs Assessment
Description: as for outcome 16
Time Frame: Baseline, week 16 and week 24
Population: As-treated population
Measure: Mean (Standard Deviation); unit: Pulse Rate (beats/min)
Arm/Group | Placebo | MEDI3506 Dose 1 | MEDI3506 Dose 2 | MEDI3506 Dose 3
Number analyzed (Participants) | 56 | 19 | 18 | 55
Pulse Rate (beats/min)
  Baseline | 68.1 (9.8) | 66.6 (8.7) | 71.3 (9.3) | 68.2 (11.1)
  Week 16: number analyzed (Participants) | 56 | 15 | 13 | 42
  Week 16 | 69.4 (10.1) | 66.9 (10.6) | 65.9 (8.6) | 66.4 (11.0)
  Week 24: number analyzed (Participants) | 56 | 16 | 13 | 40
  Week 24 | 72.0 (13.5) | 67.0 (10.4) | 74.1 (8.7) | 67.6 (10.1)

19. Secondary Outcome: Respiratory Rate Collected During Vital Signs Assessment
Description: as for outcome 16
Time Frame: Baseline, week 16 and week 24
Population: As-treated population
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Placebo | MEDI3506 Dose 1 | MEDI3506 Dose 2 | MEDI3506 Dose 3
Number analyzed (Participants) | 56 | 19 | 18 | 55
breaths/min
  Baseline | 15.4 (2.2) | 16.0 (1.5) | 16.2 (1.8) | 15.5 (1.8)
  Week 16: number analyzed (Participants) | 56 | 15 | 13 | 42
  Week 16 | 16.0 (2.3) | 15.7 (1.8) | 16.3 (1.9) | 15.9 (1.4)
  Week 24: number analyzed (Participants) | 56 | 16 | 13 | 40
  Week 24 | 15.8 (2.4) | 16.1 (1.5) | 17.1 (2.4) | 15.6 (1.6)

20. Secondary Outcome: Number of Participants With Abnormal Laboratory Assessments Relative to Normal Ranges for Haematology
Description: To assess the safety and tolerability of MEDI3506 compared with placebo, in adult subjects with moderate-to-severe AD.
Time Frame: up to 24 weeks
Population: As-treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI3506 Dose 1 | MEDI3506 Dose 2 | MEDI3506 Dose 3
Number analyzed (Participants) | 56 | 19 | 18 | 55
Participants
  Basophils: At Least One Post-Baseline Value Below LLN | 0 | 0 | 0 | 0
  Basophils: At Least One Post-Baseline Value Above ULN | 3 | 0 | 0 | 0
  Basophils: Values within normal range | 53 | 19 | 18 | 55
  Eosinophils: At Least One Post-Baseline Value Below LLN | 0 | 0 | 0 | 0
  Eosinophils: At Least One Post-Baseline Value Above ULN | 22 | 4 | 5 | 14
  Eosinophils: Values within normal range | 34 | 15 | 13 | 41
  Hematocrit: At Least One Post-Baseline Value Below LLN | 4 | 3 | 2 | 7
  Hematocrit: At Least One Post-Baseline Value Above ULN | 0 | 0 | 1 | 0
  Hematocrit: Values within normal range | 52 | 16 | 15 | 48
  Haemoglobin: At Least One Post-Baseline Value Below LLN | 5 | 1 | 3 | 8
  Haemoglobin: At Least One Post-Baseline Value Above ULN | 0 | 0 | 1 | 0
  Haemoglobin: Values within normal range | 51 | 18 | 14 | 47
  Lymphocytes: At Least One Post-Baseline Value Below LLN | 6 | 0 | 3 | 10
  Lymphocytes: At Least One Post-Baseline Value Above ULN | 0 | 0 | 0 | 0
  Lymphocytes: Values within normal range | 50 | 19 | 15 | 45
  Monocytes: At Least One Post-Baseline Value Below LLN | 1 | 0 | 1 | 3
  Monocytes: At Least One Post-Baseline Value Above ULN | 2 | 0 | 2 | 3
  Monocytes: Values within normal range | 53 | 19 | 15 | 49
  Platelet count: At Least One Post-Baseline Value Below LLN | 1 | 1 | 0 | 0
  Platelet count: At Least One Post-Baseline Value Above ULN | 3 | 0 | 2 | 5
  Platelet count: Values within normal range | 52 | 18 | 16 | 50
  Erythrocytes: At Least One Post-Baseline Value Below LLN | 10 | 3 | 4 | 17
  Erythrocytes: At Least One Post-Baseline Value Above ULN | 0 | 0 | 0 | 0
  Erythrocytes: Values within normal range | 46 | 16 | 14 | 38
  White blood cell count: At Least One Post-Baseline Value Below LLN | 7 | 1 | 2 | 6
  White blood cell count: At Least One Post-Baseline Value Above ULN | 5 | 2 | 0 | 2
  White blood cell count: Values within normal range | 44 | 16 | 16 | 47

21. Secondary Outcome: Number of Participants With Abnormal Laboratory Assessments Relative to Normal Ranges for Serum Chemistry
Description: To assess the safety and tolerability of MEDI3506 compared with placebo, in adult subjects with moderate-to-severe AD.
Time Frame: up to 24 weeks
Population: As-treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI3506 Dose 1 | MEDI3506 Dose 2 | MEDI3506 Dose 3
Number analyzed (Participants) | 56 | 19 | 18 | 55
Participants
  Albumin: At Least One Post-Baseline Value Below LLN | 0 | 0 | 0 | 0
  Albumin: At Least One Post-Baseline Value Above ULN | 21 | 5 | 6 | 15
  Albumin: Values within normal range | 35 | 14 | 12 | 40
  Alkaline Phosphatase: At Least One Post-Baseline Value Below LLN | 3 | 0 | 0 | 2
  Alkaline Phosphatase: At Least One Post-Baseline Value Above ULN | 3 | 2 | 2 | 4
  Alkaline Phosphatase: Values within normal range | 50 | 17 | 16 | 49
  Alanine Aminotransferase: At Least One Post-Baseline Value Below LLN | 0 | 0 | 0 | 0
  Alanine Aminotransferase: At Least One Post-Baseline Value Above ULN | 7 | 4 | 4 | 5
  Alanine Aminotransferase: Values within normal range | 49 | 15 | 14 | 50
  Aspartate Aminotransferase: At Least One Post-Baseline Value Below LLN | 0 | 0 | 0 | 0
  Aspartate Aminotransferase: At Least One Post-Baseline Value Above ULN | 6 | 3 | 3 | 8
  Aspartate Aminotransferase: Values within normal range | 50 | 16 | 15 | 47
  Bilirubin: At Least One Post-Baseline Value Below LLN | 0 | 0 | 0 | 0
  Bilirubin: At Least One Post-Baseline Value Above ULN | 3 | 0 | 1 | 1
  Bilirubin: Values within normal range | 53 | 19 | 17 | 54
  Urea Nitrogen: At Least One Post-Baseline Value Below LLN | 0 | 0 | 0 | 0
  Urea Nitrogen: At Least One Post-Baseline Value Above ULN | 0 | 0 | 0 | 2
  Urea Nitrogen: Values within normal range | 56 | 19 | 18 | 53
  Creatinine: At Least One Post-Baseline Value Below LLN | 0 | 0 | 0 | 0
  Creatinine: At Least One Post-Baseline Value Above ULN | 0 | 0 | 1 | 3
  Creatinine: Values within normal range | 56 | 19 | 17 | 52
  Gamma Glutamyl Transferase: At Least One Post-Baseline Value Below LLN | 4 | 2 | 0 | 5
  Gamma Glutamyl Transferase: At Least One Post-Baseline Value Above ULN | 2 | 3 | 2 | 1
  Gamma Glutamyl Transferase: Values within normal range | 50 | 14 | 16 | 49
  Potassium: At Least One Post-Baseline Value Below LLN | 1 | 1 | 0 | 1
  Potassium: At Least One Post-Baseline Value Above ULN | 1 | 0 | 1 | 1
  Potassium: Values within normal range | 54 | 18 | 17 | 53
  Sodium: At Least One Post-Baseline Value Below LLN | 0 | 0 | 0 | 0
  Sodium: At Least One Post-Baseline Value Above ULN | 2 | 0 | 0 | 2
  Sodium: Values within normal range | 54 | 19 | 18 | 53

22. Secondary Outcome: Number of Participants With Abnormal Laboratory Assessments Relative to Normal Ranges for Urinalysis
Description: To assess the safety and tolerability of MEDI3506 compared with placebo, in adult subjects with moderate-to-severe AD.
Time Frame: up to 24 weeks
Population: As-treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI3506 Dose 1 | MEDI3506 Dose 2 | MEDI3506 Dose 3
Number analyzed (Participants) | 56 | 19 | 18 | 55
Participants
  pH: At Least One Post-Baseline Value Below LLN | 0 | 0 | 0 | 0
  pH: At Least One Post-Baseline Value Above ULN | 0 | 0 | 0 | 1
  pH: Values within normal range | 56 | 19 | 18 | 54
  Erythrocytes: At Least One Post-Baseline Value Below LLN | 0 | 0 | 0 | 0
  Erythrocytes: At Least One Post-Baseline Value Above ULN | 8 | 2 | 1 | 6
  Erythrocytes: Values within normal range | 48 | 17 | 17 | 49
  Specific gravity: At Least One Post-Baseline Value Below LLN | 0 | 0 | 0 | 0
  Specific gravity: At Least One Post-Baseline Value Above ULN | 4 | 0 | 3 | 7
  Specific gravity: Values within normal range | 52 | 19 | 15 | 48
  Leukocytes: At Least One Post-Baseline Value Below LLN | 0 | 0 | 0 | 0
  Leukocytes: At Least One Post-Baseline Value Above ULN | 4 | 2 | 1 | 5
  Leukocytes: Values within normal range | 52 | 17 | 17 | 50

23. Secondary Outcome: Heart Rate (Beats/Min) Recorded on ECGs
Description: Collectively with other ECG parameters are used t assess the safety and tolerability of MEDI3506 compared with placebo, in adult subjects with moderate-to-severe AD.
Time Frame: Baseline, week 16 and week 24
Population: As-treated population
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | MEDI3506 Dose 1 | MEDI3506 Dose 2 | MEDI3506 Dose 3
Number analyzed (Participants) | 56 | 19 | 18 | 55
beats per minute
  Baseline | 67.59 (9.82) | 65.61 (6.87) | 72.63 (9.82) | 65.18 (9.43)
  Week 16: number analyzed (Participants) | 56 | 15 | 12 | 42
  Week 16 | 66.02 (9.97) | 63.80 (8.56) | 65.42 (9.08) | 63.05 (10.61)
  Week 24: number analyzed (Participants) | 56 | 16 | 13 | 40
  Week 24 | 68.17 (13.94) | 63.88 (10.41) | 72.46 (9.12) | 64.58 (9.43)

24. Secondary Outcome: QT (Miliseconds) Recorded on ECGs
Description: Collectively with other ECG parameters are used to assess the safety and tolerability of MEDI3506 compared with placebo, in adult subjects with moderate-to-severe AD.
Time Frame: Baseline, week 16 and week 24
Population: As-treated population
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | MEDI3506 Dose 1 | MEDI3506 Dose 2 | MEDI3506 Dose 3
Number analyzed (Participants) | 56 | 19 | 18 | 55
milliseconds
  Baseline | 385.43 (27.75) | 390.67 (20.57) | 380.04 (26.38) | 390.27 (22.69)
  Week 16: number analyzed (Participants) | 56 | 15 | 12 | 42
  Week 16 | 387.05 (26.14) | 390.40 (24.24) | 395.75 (20.36) | 391.95 (29.22)
  Week 24: number analyzed (Participants) | 56 | 16 | 13 | 40
  Week 24 | 385.88 (34.31) | 398.69 (28.52) | 383.15 (19.05) | 393.40 (26.54)

25. Secondary Outcome: Number of Participants With Investigator's Overall ECGs Evaluations, e.g. Normal/Abnormal and Their Clinical Significance
Description: as for outcome 24
Time Frame: Week 16 and week 24
Population: As-treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI3506 Dose 1 | MEDI3506 Dose 2 | MEDI3506 Dose 3
Number analyzed (Participants) | 56 | 19 | 18 | 55
Participants
  Week 16: Abnormal ECG: Clinically significant | 0 | 0 | 0 | 0
  Week 16: Abnormal ECG: Not Clinically significant | 3 | 2 | 2 | 10
  Week 16: Normal ECG | 38 | 13 | 10 | 32
  Week 16: Missing | 15 | 4 | 6 | 13
  Week 24: Abnormal ECG: Clinically significant | 0 | 0 | 0 | 0
  Week 24: Abnormal ECG: Not Clinically significant | 4 | 4 | 2 | 11
  Week 24: Normal ECG | 38 | 12 | 11 | 29
  Week 24: Missing | 14 | 3 | 5 | 15

26. Secondary Outcome: Left Ventricular Ejection Fraction Measured by Echocardiogram
Description: To assess the safety and tolerability of MEDI3506 compared with placebo, in adult subjects with moderate-to-severe AD.
Time Frame: Baseline and week 16
Population: As-treated population
Measure: Mean (Standard Deviation); unit: % LVEF
Arm/Group | Placebo | MEDI3506 Dose 1 | MEDI3506 Dose 2 | MEDI3506 Dose 3
Number analyzed (Participants) | 56 | 19 | 18 | 55
% LVEF
  Baseline | 64.3 (6.3) | 64.7 (6.2) | 62.8 (5.2) | 63.6 (4.7)
  Week 16: number analyzed (Participants) | 56 | 14 | 3 | 19
  Week 16 | 64.3 (5.9) | 63.0 (4.4) | 61.0 (3.6) | 65.2 (5.1)

27. Secondary Outcome: Serum MEDI3506 Concentration Profiles
Description: To evaluate the PK of MEDI3506 in adult subjects with moderate-to-severe AD.
Time Frame: Week 16 and week 24
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | MEDI3506 Dose 1 | MEDI3506 Dose 2 | MEDI3506 Dose 3
Number analyzed (Participants) | 18 | 17 | 48
μg/mL
  Week 16: number analyzed (Participants) | 15 | 14 | 33
  Week 16 | 0.377 (242) | 2.158 (193) | 5.979 (118)
  Week 24: number analyzed (Participants) | 16 | 13 | 32
  Week 24 | 0.018 (184) | 0.118 (298) | 0.188 (234)

28. Secondary Outcome: Occurence of Anti-drug Antibody During the Treatment and Follow-up Periods
Description: To evaluate the immunogenicity of MEDI3506 in adult subjects with moderate-to-severe AD.
Time Frame: up to 24 weeks
Population: As-treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI3506 Dose 1 | MEDI3506 Dose 2 | MEDI3506 Dose 3
Number analyzed (Participants) | 56 | 19 | 18 | 55
Participants
  Baseline ADA result: number analyzed (Participants) | 55 | 19 | 18 | 53
  Baseline ADA result | 1 | 0 | 0 | 0
  Post-baseline ADA result | 1 | 1 | 0 | 2

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Placebo | MEDI3506 Dose 1 | MEDI3506 Dose 2 | MEDI3506 Dose 3
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/19 | 0/18 | 0/55
Serious Adverse Events (participants affected / at risk) | 2/56 | 0/19 | 2/18 | 1/55
Other Adverse Events (participants affected / at risk) | 29/56 | 11/19 | 14/18 | 25/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=56) | MEDI3506 Dose 1 (N=19) | MEDI3506 Dose 2 (N=18) | MEDI3506 Dose 3 (N=55)
Food allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=56) | MEDI3506 Dose 1 (N=19) | MEDI3506 Dose 2 (N=18) | MEDI3506 Dose 3 (N=55)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (6)
Injection site swelling (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 7 (7) | 0 (0) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis infected (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema infected (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Urine analysis abnormal (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 12 (14) | 2 (2) | 0 (0) | 14 (17)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 2 (2) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/69/NCT04212169/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-08): https://cdn.clinicaltrials.gov/large-docs/69/NCT04212169/SAP_001.pdf